CLINICAL TRIAL: NCT05613894
Title: A Phase Ib Dose-Escalation Study of Cabozantinib in Combination With Lutetium-177 (177Lu)-PSMA-617 in Patients With Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Brief Title: Dose-Escalation Study of Cabozantinib in Combination With Lutetium-177 (177Lu)-PSMA-617 in Patients With Metastatic Castration-Resistant Prostate Cancer
Acronym: CaboLu
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HCI157278
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
MeSH Terms: interventions — cabozantinib; Pluvicto

STUDY DESIGN:
Intervention Model Description: A standard 3+3 dose escalation design will be used to identify the MTD and/or recommended dose and schedule for the subsequent expansion phase. The study will test 2 dose levels of cabozantinib with the option to dose reduce to dose level -1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Part 1) (Experimental): Part 1 will assess the rate of dose-limiting toxicities (DLTs) during the DLT evaluation period and identify the MTD and/or recommended dose and schedule
  Interventions: Drug: Cabozantinib
- Dose Expansion Cohort (Part 2) (Experimental): Expansion Phase to assess identified MTD and schedule from Part 1.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — (177Lu)-PSMA-617 will be administered every 6 weeks for up to 6 cycles per SOC. Oral Cabozantinib taken daily at home.
  Other Names: 177Lu-PSMA-617

SUMMARY:
This is an open-label, phase 1b dose-escalation study of cabozantinib in combination with 177Lu-PSMA-617 in subjects with mCRPC. The primary hypothesis is that cabozantinib with 177Lu-PSMA will be safe and have efficacy in patients with mCRPC. The dose-escalation phase (Part 1) will assess the rate of dose-limiting toxicities (DLTs) during the DLT evaluation period and identify the MTD and/or recommended dose and schedule for the subsequent expansion phase (Part 2).

ELIGIBILITY:
Inclusion Criteria:

* Male subject aged ≥ 18 years.
* Histologically or cytologically confirmed adenocarcinoma of the prostate without small cell histology.
* Prior orchiectomy and/or ongoing androgen-deprivation therapy and a castrate level of serum testosterone (<50 ng/dL or <1.7 nmol/L).
* Prior treatment with at least one prior Novel Hormone Therapy (NHT), defined as second-generation anti-androgen therapies that include, but are not limited to, abiraterone acetate, enzalutamide, apalutamide, and darolutamide.
* Must be eligible for therapy with 177Lu-PSMA-617 and have ≥ 1 PSMA-positive lesion per treating investigator.
* Must have progressive mCRPC per the treating investigator.
* ECOG Performance Status ≤ 1.
* Adequate organ function as defined as:

  * Hematologic:

    * Absolute neutrophil count (ANC) ≥ 1500/µL without granulocyte colony-stimulating factor support
    * White blood cell count ≥ 3000/µL.
    * Platelet count ≥ 100,000/µL
    * Hemoglobin ≥ 9g/dL
    * Serum albumin ≥ 2.5 g/dl
    * PT/INR or partial thromboplastin time (PTT) test < 1.3x the laboratory ULN
  * Hepatic:

    * Total Bilirubin ≤ 1.5x institutional upper limit of normal (ULN)
    * For subjects with Gilbert's disease: ≤ 3x ULN
    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3x upper limit of normal (ULN).
  * Renal:

    * Urine protein/creatinine ratio (UPCR) ≤ 1 mg/mg (≤ 113.2 mg/mmol), or 24-h urine protein ≤ 1 g
    * Estimated creatinine clearance ≥ 50 mL/min by Cockcroft-Gault formula Males: ((140-age)×weight[kg])/(serum creatinine [mg/dL]×72)
* Sexually active fertile patients and their partners must agree to use medically accepted methods of contraception (e.g., barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 6 months after the last dose of study treatment in accordance with section 5.4.2.
* Recovery to baseline or ≤ Grade 1 CTCAE v5 from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.
* Patients must have a life expectancy >3 months.

Exclusion Criteria:

* Receiving other investigational anti-cancer agents.
* Prior treatment with cabozantinib
* Previous treatment with Strontium-89, Samarium-153, Rhenium-186, Rhenium-188, Radium-223 or hemi-body irradiation within 6 months prior to randomization.
* Previous PSMA-targeted radioligand therapy
* Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 2 weeks before first dose of study treatment.
* Receipt of any type of cytotoxic, biologic or other systemic anticancer therapy (including investigational) within 4 weeks before first dose of study treatment.
* Radiation therapy for bone metastasis within 2 weeks or any other radiation therapy within 4 weeks before first dose of study treatment.
* Systemic treatment with radionuclides within 6 weeks before first dose of study treatment.
* Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.
* Symptomatic cord compression, or clinical or radiologic findings indicative of impending cord compression.
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks prior to first dose of study treatment after radiotherapy or at least 4 weeks prior to first dose of study treatment after major surgery (e.g., removal or biopsy of brain metastasis).
* Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment.
* Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of first dose of study treatment.
* Major surgery within 4 weeks prior to starting study drug, minor surgery within 10 days, or subjects who have not fully recovered from major surgery.
* Any other active malignancy at time of first dose of study treatment or diagnosis of another malignancy within 3 years prior to first dose of study treatment that requires active treatment, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%), such as locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the breast.
* Concomitant anticoagulation with coumarin agents (e.g., warfarin), direct thrombin inhibitors (e.g., dabigatran), direct factor Xa inhibitor betrixaban, or platelet inhibitors (e.g., clopidogrel). Allowed anticoagulants are the following:

  * Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH)
  * Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor.
* Current evidence of uncontrolled, significant intercurrent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders:

    * Congestive heart failure New York Heart Association Class III or IV, unstable angina pectoris, serious cardiac arrhythmias.
    * Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic events, or thromboembolic event (eg, deep venous thrombosis, pulmonary embolism) within 6 months before the first dose of study treatment.
    * Subjects with a diagnosis of incidental, subsegmental PE or DVT within 6 months are allowed if stable, asymptomatic, and treated with a stable dose of permitted anticoagulation (see exclusion criterion 14) for at least 1 week before first dose of study treatment.
    * Uncontrolled hypertension defined as sustained blood pressure (BP) ≥ 150 mm Hg systolic or >90 mmHg diastolic despite optimal antihypertensive treatment.
  * Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:

    * The subject has evidence of tumor invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (e.g., Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction.
    * Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose of study treatment.
    * Note: Complete healing of an intra-abdominal abscess must be confirmed before first dose of study treatment.
  * Any other condition that would, in the Investigator's judgment, contraindicate the subject's participation in the clinical study due to safety concerns or compliance with clinical study procedures (e.g., infection/inflammation, intestinal obstruction, unable to swallow medication, social/ psychological issues, etc.)
* Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (e.g., pulmonary hemorrhage) within 12 weeks before first dose of study treatment.
* Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation.
* Lesions invading or encasing any major blood vessels
* Other clinically significant disorders that would preclude safe study participation.

  * Serious non-healing wound/ulcer/bone fracture.
  * Uncompensated/symptomatic hypothyroidism.
  * Moderate to severe hepatic impairment (Child-Pugh B or C).
  * Known history of COVID-19 unless the subject has clinically recovered from the disease at least 30 days prior to first dose of study treatment.
* Major surgery (e.g., laparoscopic nephrectomy, GI surgery, removal or biopsy of brain metastasis) within 2 weeks before first dose of study treatment or minor surgeries within 10 days before first dose of study treatment.
* Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment.

  --Subjects with clinically relevant ongoing complications from prior surgery are not eligible.
* Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms per electrocardiogram (ECG) within 28 days before first dose of study treatment.

  --Note: If a single ECG shows a QTcF with an absolute value > 500 ms, two additional ECGs at intervals of approximately 3 min must be performed within 30 min after the initial ECG, and the average of these three consecutive results for QTcF will be used to determine eligibility.
* Inability to swallow tablets
* Previously identified allergy or hypersensitivity to components of the study treatment formulations.
* Known HIV infection with a detectable viral load within 6 months of the anticipated start of treatment.

  --Note: Subjects on effective antiretroviral therapy with an undetectable viral load within 6 months of the anticipated start of treatment are eligible for this trial.
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination, radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), or hepatitis C.
* Note: Subjects with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Subjects positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Medical, psychiatric, cognitive, or other conditions that may compromise the subject's ability to understand the subject information, give informed consent, comply with the study protocol or complete the study.
* Subjects taking prohibited medications as described in Section 6.8.2. A washout period of prohibited medications for a period of at least five half-lives or as clinically indicated should occur before the start of treatment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male
Enrollment: 33 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
The rate of dose-limiting toxicities (DLTs) during the DLT evaluation period | 28 days
  To determine the maximum tolerated dose (MTD) and recommended dose and schedule for the subsequent Expansion Stage of daily oral administration of cabozantinib in subjects with metastatic castration-resistant prostate cancer (mCRPC) when taken in combination with 177Lu-PSMA-617
The proportion of patients without progression as defined by PCWG3-modified RECIST 1.1 at 24 weeks. | 24 weeks
  To evaluate preliminary efficacy by estimating the progression-free survival (PFS) at 24 weeks (PFS24w) as assessed by per PCWG3-modified RECIST v1.1

SECONDARY OUTCOMES:
The frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by type, severity (as defined by the NCI CTCAE, version 5.0), seriousness, duration, and relationship to study treatment. | up to 2 years
  To assess the safety and tolerability of 177Lu-PSMA and cabozantinib in the study population
ORR, defined as the proportion of subjects with measurable disease achieving a confirmed PR and CR as defined by PCWG3-modified RECIST 1.1. | 3 years
  To assess the objective response rate (ORR) in the study population.
DoR, defined as the interval of time from the date of initial documented response (PR or better per PCWG3-modified RECIST 1.1) to the time of progression from the best response, the start of a new therapy, or death from any cause. | up to 3 years
  To assess the duration of response (DoR) of the study population.
rPFS as assessed by PCWG3-modified RECIST 1.1 from start of therapy to the time of radiographic progression or death from any cause. | up to 3 years
  To assess the radiographic PFS (rPFS) of the study population.
The proportion of patients without progression as defined by PCWG3-modified RECIST 1.1 at 38 weeks. | 38 weeks
  To evaluate PFS at 38 weeks (PFS38w) as assessed by per PCWG3-modified RECIST v1.1.
The levels of PSA will be monitored every 3 (or 4) weeks for comparison to baseline levels until the time of PSA progression, as defined by PCWG3 criteria. | 4 weeks
  To assess the PSA PFS of the study population.
The levels of PSA will be monitored per treatment schedule to assess the proportion of patients with a 50% reduction in PSA levels (PSA50) compared to the baseline value at the time of study enrollment. | up to 2 years
  To assess the PSA 50% response rate in the study population.
OS as defined as the time from registration until death from any cause. | up to 3 years
  To assess overall survival (OS) in this study population

CONTACTS AND LOCATIONS:
Overall Officials: Umang Swami, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No